CLINICAL TRIAL: NCT07125781
Title: Prevalence of Central Sensitization and Nociplastic Pain in Individuals Diagnosed With Pes Planus: A Multicenter Cross-Sectional Study
Brief Title: Central Sensitization and Nociplastic Pain in Pes Planus
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Other Study IDs: 2024/30
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pes Planus; Flatfoot; Central Sensitization; Nociplastic Pain
Keywords: Pes Planus; Flatfoot; Central Sensitization Inventory; Nociplastic Pain; Pain-DETECT Questionnaire; Foot Function Index; Chronic Foot Pain; Biopsychosocial Pain Mechanisms
MeSH Terms: conditions — Flatfoot; Nociplastic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the patient group: Adults aged 18 to 65 years with a clinical diagnosis of pes planus confirmed by a physical medicine and rehabilitation specialist, experiencing lower extremity pain for at least six months. Participants completed validated questionnaires to assess pain intensity, foot function, nociplastic pain features, central sensitization, psychological status, and quality of life. No therapeutic intervention was administered as part of the study.
- The control group: Age- and sex-matched healthy volunteers with no current or past foot or leg pain. Participants had no history of pes planus, lower limb surgery, trauma, or rheumatologic, neurologic, endocrine, or vascular disorders that could influence pain perception. No interventions were applied; they completed the same validated questionnaires as the pes planus group for comparison purposes.

SUMMARY:
Background:

Pes planus, commonly known as flatfoot, is a condition characterized by the collapse of the medial longitudinal arch of the foot. While some individuals remain asymptomatic, many experience foot or leg pain, walking difficulties, and functional limitations. In some cases, symptoms persist despite adequate conventional treatment. This suggests that central pain mechanisms, such as central sensitization and nociplastic pain, may contribute to ongoing symptoms. These mechanisms involve changes in the central nervous system that amplify pain perception and can occur even in the absence of active tissue damage. Understanding these mechanisms in pes planus may help guide more targeted and effective treatment strategies.

Purpose:

The aim of this multicenter cross-sectional study was to determine the prevalence of central sensitization and nociplastic pain in individuals with clinically diagnosed pes planus and to compare the findings with age- and sex-matched healthy controls.

Methods:

Between November 2024 and May 2025, a total of 107 patients with pes planus and 107 healthy controls were recruited from three medical centers. Participants completed validated Turkish versions of the Visual Analog Scale for pain intensity, the Foot Function Index for functional limitation, the Pain-DETECT questionnaire for nociplastic pain symptoms, the Central Sensitization Inventory for central sensitization, the Hospital Anxiety and Depression Scale for psychological distress, and the Short Form-12 for quality of life. Data were analyzed using comparative statistical tests and multiple linear regression models to identify factors associated with nociplastic pain and central sensitization in the pes planus group.

DETAILED DESCRIPTION:
Pes planus, also referred to as flatfoot, is a common musculoskeletal condition characterized by the flattening or collapse of the medial longitudinal arch of the foot. It affects a considerable portion of the adult population and may be associated with foot pain, functional impairment, and reduced quality of life. In many patients, pain symptoms persist despite adequate structural correction and conventional treatments such as footwear modifications, orthotic support, exercise, or anti-inflammatory medications. This persistence suggests that central mechanisms of pain processing may be involved.

Central sensitization is a phenomenon in which the central nervous system exhibits heightened responsiveness to sensory input, resulting in amplified pain perception even in the absence of ongoing tissue injury. Nociplastic pain is a relatively new classification describing pain arising from altered central nociceptive processing without clear evidence of tissue damage or nerve injury. Both mechanisms are increasingly recognized in chronic musculoskeletal disorders, yet they have been underexplored in individuals with pes planus.

This multicenter cross-sectional study was designed to investigate the prevalence of central sensitization and nociplastic pain in adults with clinically diagnosed pes planus and to compare these findings with healthy controls matched for age and sex. Participants were recruited from three medical centers between November 2024 and May 2025. Inclusion criteria required adults aged 18 to 65 years with lower extremity pain lasting at least six months and a diagnosis of pes planus confirmed by a physical medicine and rehabilitation specialist. Healthy controls had no history of foot or leg pain or relevant musculoskeletal disorders.

All participants completed standardized and validated assessment tools, including the Visual Analog Scale for pain intensity, the Foot Function Index for foot-related disability, the Pain-DETECT questionnaire for nociplastic pain features, the Central Sensitization Inventory for signs of central sensitization, the Hospital Anxiety and Depression Scale for psychological distress, and the Short Form-12 for quality of life. Demographic and clinical information was also recorded.

Statistical analyses compared results between the pes planus and control groups and examined correlations among pain severity, functional impairment, central sensitization, nociplastic pain, and psychological measures. Multiple linear regression models were used to identify independent predictors of nociplastic pain and central sensitization in the pes planus group.

The findings of this study are intended to improve understanding of the complex pain mechanisms associated with pes planus and to highlight the potential need for multidisciplinary management approaches that address central pain processes and psychological factors alongside conventional biomechanical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* For pes planus group: clinically diagnosed pes planus confirmed by physical medicine and rehabilitation specialists, with persistent lower extremity pain for at least 6 months.
* For control group: age- and sex-matched healthy volunteers without current or past foot or leg pain.
* Willingness to complete all self-report questionnaires.
* Provided written and verbal informed consent.

Exclusion Criteria:

* History of diabetes mellitus, hypothyroidism, malignancy, vasculitis, neuropathies, or lumbar radiculopathy.
* History of lower limb surgery or trauma.
* Recent local injection or extracorporeal shockwave therapy.
* Any rheumatologic disease affecting pain perception (e.g., rheumatoid arthritis, ankylosing spondylitis).
* Severe psychiatric disorder or cognitive impairment interfering with questionnaire completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years, including individuals with clinically diagnosed pes planus and age- and sex-matched healthy volunteers without lower extremity pain. Participants were recruited from physical medicine and rehabilitation clinics at Etlik Zübeyde Hanım Gynecology and Pediatrics Training and Research Hospital, Ankara Etlik City Hospital, and Yozgat City Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Pain-DETECT questionnaire | Baseline
  The Pain-DETECT questionnaire consists of 9 items with a total score range of 1-38. Scores ≤12 indicate that neuropathic or nociplastic pain components are unlikely, 13-18 indicate uncertainty, and ≥19 indicate probable nociplastic or neuropathic pain. The validated Turkish version, developed by Alkan et al. (2013), demonstrated a sensitivity of 90% and specificity of 67.5% for the ≤12 cutoff, with a negative predictive value of 87%.
Central Sensitization Inventory | Baseline
  The Central Sensitization Inventory contains 25 items scored 0-4 (0 = never, 4 = always). Total scores ≥40 indicate the presence of central sensitization, with severity categories as follows: 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, ≥60 very severe. The validated Turkish version, developed by Keleş et al. (2021), reported 81% sensitivity and 75% specificity for the ≥40 cutoff, with excellent internal consistency (Cronbach's alpha = 0.92) and test-retest reliability (intraclass correlation coefficient = 0.93).

SECONDARY OUTCOMES:
Visual Analog Scale | Baseline
  The Visual Analog Scale is a 10 cm horizontal line anchored with "0 = no pain" and "10 = very severe pain." Participants mark their pain severity at rest and during activity for each foot. Higher scores indicate greater pain intensity.
Foot Function Index | Baseline
  The Foot Function Index consists of 23 items across three subscales: pain (9 items), disability (9 items), and activity limitation (5 items). Each item is scored using a 10 cm visual analog scale reflecting the previous week's foot condition. Higher scores indicate greater impairment. The Turkish version was adapted and validated by Yalıman et al., with cultural and linguistic modifications for plantar fasciitis patients.
Hospital Anxiety and Depression Scale | Baseline
  The Hospital Anxiety and Depression Scale contains 14 items, split evenly into anxiety and depression subscales, each scored 0-21. Interpretation: 0-7 = normal, 8-10 = mild, 11-14 = moderate, 15-21 = severe. The validated Turkish version was developed by Aydemir et al. (1997).
Short Form-12 Health Survey (SF-12) | Baseline
  The Short Form-12 assesses physical and mental components of health-related quality of life across eight domains. Higher scores indicate better quality of life. The validated Turkish version was established in 2022 by Soylu and Kütük.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article (after deidentification) will be made available upon reasonable request to the corresponding author after publication. Data will be shared with researchers who provide a methodologically sound proposal for use in achieving the aims stated in their proposal. Requests should be directed to gulserendmr58@hotmail.com. Data will be available for 12 months following article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting materials will be available beginning 6 months after publication of the main study results and will be accessible for a period of 12 months thereafter.
Access Criteria: Data will be available to qualified researchers with a methodologically sound proposal for secondary analyses related to the study objectives. Requests should be submitted to the corresponding author at gulserendmr58@hotmail.com. Approved requestors will be provided access via secure email or institutional file transfer systems.
URL: http://tip.bozok.edu.tr

REFERENCES:
- [Background] Alkan H, Ardic F, Erdogan C, Sahin F, Sarsan A, Findikoglu G. Turkish version of the painDETECT questionnaire in the assessment of neuropathic pain: a validity and reliability study. Pain Med. 2013 Dec;14(12):1933-43. doi: 10.1111/pme.12222. Epub 2013 Aug 7. PMID 23924395
- [Background] Buldys K, Gornicki T, Kalka D, Szuster E, Biernikiewicz M, Markuszewski L, Sobieszczanska M. What Do We Know about Nociplastic Pain? Healthcare (Basel). 2023 Jun 17;11(12):1794. doi: 10.3390/healthcare11121794. PMID 37372912